CLINICAL TRIAL: NCT06748690
Title: Comparison of Endoscopic Mucosal Cutting Biopsy and Endoscopic Ultrasound-guided-fine Needle Aspiration for Preoperative Pathological Evaluation of Gastric Submucosal Tumors
Brief Title: MCB vs EUS-FNA for Preoperative Pathological Evaluation of Gastric SMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Liming, Director, Head of Endoscopy center, Principal Investigator, Clinical Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RDL-13
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Stromal Tumor of Stomach; Submucosal Tumor of Stomach
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCB group (Experimental): Use a disposable high-frequency cutting knife under endoscopy to cut open the surface mucosa of the tumor, and use biopsy forceps to extract tissue that can be fully evaluated for pathological examination. Use a disposable hemostatic clip to suture the mucosal incision, and after thorough observation of the hemostasis, withdraw from the endoscope.
  Interventions: Procedure: mucosal cutting biopsy
- EUS-FNA group (Active Comparator): Using standard Endoscopic Ultrasonography-Guided Fine-Needle Aspiration(EUS-FNA) technology, using endoscopic ultrasound scanning to locate lesions, and puncture needle aspiration biopsy.
  Interventions: Procedure: endoscopic ultrasound-guided-fine needle aspiration

INTERVENTIONS:
Procedure: mucosal cutting biopsy — Under intravenous anesthesia, the patient inserted a gastroscopy (Olympus GIF-260J) through the mouth and used a disposable high-frequency cutting knife to cut open the surface mucosa of the tumor. Biopsy forceps were used to extract tissue that could be fully evaluated for pathological examination. Use a disposable hemostatic clip to suture the mucosal incision, and after thorough observation of the hemostasis, withdraw from the endoscope.
  (
  Arms: MCB group
Procedure: endoscopic ultrasound-guided-fine needle aspiration — 2) EUS-FNA group: Standard (Endoscopic Ultrasonography-Guided Fine-Needle Aspiration) EUS-FNA technology was used, and electronic linear array ultrasound endoscopy (GF-UCT-260, Olympus, Japan) was used to scan and locate the lesion. Puncture needle (Boston Scientific, USA) was used for aspiration biopsy. The thickness of the puncture needle depends on the size, hardness, and location of the tumor.
  Arms: EUS-FNA group

SUMMARY:
Gastrointestinal stromal tumors (GISTs) are the most common submucosal tumors (SMTs) of the stomach. The 2022 European Society of Oncology ESMO Diagnosis and Treatment Guidelines recommend that GISTs undergo biopsy with a clear pathological diagnosis and should be removed unless there are significant complications. But currently, the diagnostic rate of EUS-FNA for upper gastrointestinal subcutaneous lesions is less than 60%. In recent years, mucosal cutting biopsy (MCB) has become an effective method for diagnosing SMTs. Regardless of whether the SMTs are large or small, the application of MCB technology can quickly obtain pathological tissue under direct visualization, and its immunohistochemical pathological diagnosis rate is relatively satisfactory. MCB technology has great potential in the biopsy of SMTs, but there is currently no comparison of results between two technologies in randomized controlled trials. The purpose of this study is to design a randomized controlled trial to compare the diagnostic rates of EUS-FNA and MCB techniques for tissue pathology (including immunohistochemistry) of SMTs, in order to improve the diagnostic accuracy of SMTs in our hospital and improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic evaluation considers gastric submucosal tumors (SMTs) with a diameter of ≥ 15mm

Exclusion Criteria:

* Endoscopic non bulging lesions.
* The upper gastrointestinal lesions measured by Endoscopic Ultrasonography(EUS) are less than 15 mm.
* Lesions that do not require tissue collection (such as lipomas, varicose veins)
* Patients with cystic lesions
* The patient has uncorrectable coagulation dysfunction (International Normalized Ratio (INR)>1.5 or platelet count<50x109)
* Patients with portal hypertension
* Patients with a history of upper gastrointestinal surgery
* Pregnant women
* Patients who refuse to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis and immunohistochemical diagnosis | Pathological evaluation should be conducted immediately after specimen isolation
  Comparison of diagnostic yield between Mucosal Cutting Biopsy (MCB) and Endoscopic Ultrasonography-Guided Fine-Needle Aspiration (EUS-FNA) The diagnostic yield was defined as the percentage of lesions confirmed by a pathologic diagnosis involving immunohistological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Liming Zhang, M.D., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhaliwal A, Kolli S, Dhindsa BS, Devani K, Ramai D, Sayles H, Rangray R, Bhat I, Singh S, Adler DG. Clinical efficacy and safety of mucosal incision-assisted biopsy for the diagnosis of upper gastrointestinal subepithelial tumors: A systematic review and meta-analysis. Ann Gastroenterol. 2020 Mar-Apr;33(2):155-161. doi: 10.20524/aog.2020.0460. Epub 2020 Feb 14. PMID 32127736
- [Background] Fernandez-Esparrach G, Sendino O, Sole M, Pellise M, Colomo L, Pardo A, Martinez-Palli G, Arguello L, Bordas JM, Llach J, Gines A. Endoscopic ultrasound-guided fine-needle aspiration and trucut biopsy in the diagnosis of gastric stromal tumors: a randomized crossover study. Endoscopy. 2010 Apr;42(4):292-9. doi: 10.1055/s-0029-1244074. Epub 2010 Mar 30. PMID 20354939
- [Background] Sanaei O, Fernandez-Esparrach G, De La Serna-Higuera C, Carrara S, Kumbhari V, El Zein MH, Ismail A, Gines A, Sendino O, Montenegro A, Repici A, Rahal D, Brewer Gutierrez OI, Moran R, Yang J, Parsa N, Paiji C, Aghaie Meybodi M, Shin EJ, Lennon AM, Kalloo AN, Singh VK, Canto MI, Khashab MA. EUS-guided 22-gauge fine needle biopsy versus single-incision with needle knife for the diagnosis of upper gastrointestinal subepithelial lesions: a randomized controlled trial. Endosc Int Open. 2020 Mar;8(3):E266-E273. doi: 10.1055/a-1075-1900. Epub 2020 Feb 21. PMID 32118100